CLINICAL TRIAL: NCT02189785
Title: Endogenous Opioid Mechanisms for Rejection Sensitivity
Status: Completed | Type: Observational
Sponsor: Stony Brook University (Other)
Collaborators: University of Michigan (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, David Hsu, Assistant Professor, Stony Brook University
Other Study IDs: R01MH102264 (NIH); R01MH102264 (NIH)
Record Dates: First submitted 2014-07-11; First posted 2014-07-15 (Estimated); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Rejection Sensitivity
Keywords: social; rejection; acceptance; PET; opioid; fMRI; reward; exclusion
MeSH Terms: conditions — Rejection, Psychology

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — saliva, whole blood, blood plasma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Healthy Controls: Healthy men and women ages 18-25 years

SUMMARY:
This project hypothesizes that the brain's opioid system determines rejection sensitivity, a personality trait that is a vulnerability factor and feature of several psychiatric disorders. This project will use positron emission tomography to measure the brain's opioid response to social rejection and acceptance in a nonclinical population with varying levels of rejection sensitivity. The results will provide the first major step towards understanding a neurotransmitter mechanism for rejection sensitivity, allowing for further investigation into predicting and treating its associated disorders.

DETAILED DESCRIPTION:
Humans depend on acceptance into groups and intimate relationships for survival and emotional well-being. Actual or perceived threats to this need such as social rejection (when one is not wanted or liked) can lead to marked changes in mood and behavior such as sadness, social withdrawal, and impulsivity. The experience of severe or repeated social rejection in those who are rejection sensitive is a strong contributor to psychiatric disorders such as major depressive, social anxiety, and personality disorders. The neurotransmitter mechanisms underlying rejection sensitivity (RS) are not known.

It has been known for over 30 years in nonhuman animals that the endogenous opioid system, particularly the µ-opioid receptor (MOR) system, regulates social distress and social reward behaviors. Using positron emission tomography, we recently showed that social rejection and acceptance produced robust MOR-mediated neurotransmission in specific brain areas, which correlated with changes in mood and behavior. This study was the first to show that the endogenous opioid system responds to social cues in humans. The proposed project will examine the MOR system in the clinically important trait of RS. Since the neurotransmitter mechanisms of RS are unknown, we seek to first understand the basic neurobiology of RS in a healthy population, prior to studying clinical populations.

The overall hypothesis is that RS is associated with MOR function. Those with higher RS compared to lower RS are hypothesized to have overall lower MOR activation during social rejection and acceptance, leading to greater distress and dampened pro-social behavior. Numerous animal studies have also established that the MOR system is strongly influenced by harmful social environments. Therefore, we will also examine the role of childhood maltreatment (CM), a negative early life experience known to be one of the highest risk factors for developing depression and anxiety. The goal of this project is to determine how RS and CM interact to determine patterns of MOR binding during baseline, social rejection, and social acceptance in a healthy population. We will also examine how RS, mediated through MOR activation, influences mood and behavior.

The impact of this research is to provide the first major step towards understanding a neurotransmitter mechanism for RS, with the long-term goal of predicting and treating its associated disorders.

ELIGIBILITY:
Inclusion Criteria:

* Men and women age 18-25 (inclusive)
* Right-handed
* Native English speaker
* Not currently in a romantic relationship
* Willing and able to participate in a PET scan

Exclusion Criteria:

* Not on hormonal birth control
* Not pregnant
* Consume less than 5 cigarettes per week and less than 14 alcoholic drinks per week, on average
* No use of recreational or street drugs in the past two years (e.g. marijuana)
* Willing to abstain from alcohol and/or tobacco for 48 hours
* No major untreated medical problems
* Never diagnosed with a psychiatric or neurological disorder
* Potential problems with having an MRI scan (claustrophobia, metal objects, etc.)

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy Controls
Sampling Method: Probability Sample
Enrollment: 114 (Actual)
Dates: Start 2016-08; Primary Completion 2019-06-06 (Actual); Study Completion 2019-06-06 (Actual)

PRIMARY OUTCOMES:
Mu-opioid binding potential | within 30 days of informed consent
  This study will measure levels of radiotracer (carbon-11-labeled carfentanil) binding to the mu-opioid receptor in the brain using positron-emission tomography (PET). Primary regions of interest include: the amygdala, anterior insular cortex, anterior cingulate cortex, nucleus accumbens, and thalamus. All structures will be examined bilaterally. Differences in binding potential (Bmax/Kd) for the radiotracer will be compared across different experimental conditions (e.g., neutral, positive, negative social feedback).

SECONDARY OUTCOMES:
fMRI blood-oxygen-level-dependent (BOLD) response | within 30 days of informed consent
  This study will measure brain activation in response to social feedback and monetary reward. Primary regions of interest include: the amygdala, anterior insular cortex, and the nucleus accumbens. All structures will be examined bilaterally. Arbitrary units for fMRI BOLD are used to compare activation during one condition (e.g., neutral, baseline) vs. another condition (e.g., positive social feedback, monetary reward).
Plasma cortisol | within 30 days of informed consent
  This study will collect blood every 10 minutes during PET to measure changes in levels of plasma cortisol. Units are ug/dL.

CONTACTS AND LOCATIONS:
Overall Officials: David T Hsu, Ph.D., Principal Investigator — Stony Brook University
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States